CLINICAL TRIAL: NCT01368289
Title: Australian Multicentre Colonic Endoscopic Mucosal Resection (ACE/EMR) Study
Brief Title: Australian Multicentre Colonic Endoscopic Mucosal Resection Study
Acronym: ACEEMR
Status: Active, not recruiting | Type: Observational
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Dr Michael Bourke, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Other Study IDs: ACE/EMR
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonic Polyps: Patients who present with colonic polyps >20mm
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection — Endoscopic Mucosal Resection of large sessile colonic polyps.

SUMMARY:
A prospective, multicentre, observational study of all patients referred for endoscopic resection of sessile colorectal polyps sized ≥20 mm conducted with intention to treat analysis.

DETAILED DESCRIPTION:
A prospective, multicentre, observational study of all patients referred for endoscopic resection of sessile colorectal polyps sized ≥20 mm conducted with intention to treat analysis. Detailed data regarding lesion characteristics (size, location, Paris classification, granular or non-granular surface morphology and Kudo pit pattern), procedural, clinical and histological outcomes and complications are noted. Multivariate analysis will be performed to identify risk factors for Endoscopic Mucosal Resection failure and adenoma recurrence at follow-up colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Large sessile polyp (equal to or greater than 20mm)
* Intention to perform EMR
* Aged 18 years or older

Exclusion Criteria:

* Colonic polyps less than 20mm
* Aged younger then 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who presents to the Unit with the intention to treat large sessile colonic polyps equal to or greater than 20mm.
Sampling Method: Probability Sample
Enrollment: 3072 (Actual)
Dates: Start 2008-09; Primary Completion 2016-11 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Technical success for Endoscopic resection | 6-60 months
  To determine the safety, efficacy and predictors of success for Endoscopic Mucosal Resection of large sessile colorectal polyps. The utility of endoscopic criteria to stratify for the risk of Submucosal Invasive Cancer was also assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, Principal Investigator — Westmead Hospital - Endoscopy Unit
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] Gauci JL, Mandarino FV, Kerrison C, Whitfield AM, O'Sullivan T, Gupta S, Lam B, Perananthan V, Cronin O, Lee EY, Williams SJ, Burgess N, Bourke MJ. Margin thermal ablation eliminates size as a risk factor for recurrence after piecemeal endoscopic mucosal resection of large non-pedunculated colorectal polyps. Gut. 2025 Apr 7;74(5):752-760. doi: 10.1136/gutjnl-2024-333563. PMID 40044497
- [Derived] Gauci JL, Whitfield A, Medas R, Kerrison C, Mandarino FV, Gibson D, O'Sullivan T, Cronin O, Gupta S, Lam B, Perananthan V, Hourigan L, Zanati S, Singh R, Raftopoulos S, Moss A, Brown G, Klein A, Desomer L, Tate DJ, Williams SJ, Lee EY, Burgess N, Bourke MJ. Prevalence of Endoscopically Curable Low-Risk Cancer Among Large (>/=20 mm) Nonpedunculated Polyps in the Right Colon. Clin Gastroenterol Hepatol. 2025 Mar;23(4):555-563.e1. doi: 10.1016/j.cgh.2024.07.017. Epub 2024 Jul 31. PMID 39089517
- [Derived] Tate DJ, Vosko S, Bar-Yishay I, Desomer L, Shahidi N, Sidhu M, McLeod D, Bourke MJ. Incomplete mucosal layer excision during EMR: a potential source of recurrent adenoma (with video). Gastrointest Endosc. 2024 Sep;100(3):501-509. doi: 10.1016/j.gie.2024.01.030. Epub 2024 Jan 25. PMID 38280532
- [Derived] Tate DJ, Desomer L, Argenziano ME, Mahajan N, Sidhu M, Vosko S, Shahidi N, Lee E, Williams SJ, Burgess NG, Bourke MJ. Treatment of adenoma recurrence after endoscopic mucosal resection. Gut. 2023 Oct;72(10):1875-1886. doi: 10.1136/gutjnl-2023-330300. Epub 2023 Jul 6. PMID 37414440
- [Derived] Gupta S, Vosko S, Shahidi N, O'Sullivan T, Cronin O, Whitfield A, Kurup R, Sidhu M, Lee EYT, Williams SJ, Burgess NG, Bourke MJ. Endoscopic resection-related colorectal strictures: risk factors, management, and long-term outcomes. Endoscopy. 2023 Nov;55(11):1010-1018. doi: 10.1055/a-2106-6494. Epub 2023 Jun 6. PMID 37279786
- [Derived] O'Sullivan T, Tate D, Sidhu M, Gupta S, Elhindi J, Byth K, Cronin O, Whitfield A, Craciun A, Singh R, Brown G, Raftopoulos S, Hourigan L, Moss A, Klein A, Heitman S, Williams S, Lee E, Burgess NG, Bourke MJ. The Surface Morphology of Large Nonpedunculated Colonic Polyps Predicts Synchronous Large Lesions. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2270-2277.e1. doi: 10.1016/j.cgh.2023.01.034. Epub 2023 Feb 12. PMID 36787836
- [Derived] Cronin O, Sidhu M, Shahidi N, Gupta S, O'Sullivan T, Whitfield A, Wang H, Kumar P, Hourigan LF, Byth K, Burgess NG, Bourke MJ. Comparison of the morphology and histopathology of large nonpedunculated colorectal polyps in the rectum and colon: implications for endoscopic treatment. Gastrointest Endosc. 2022 Jul;96(1):118-124. doi: 10.1016/j.gie.2022.02.022. Epub 2022 Feb 24. PMID 35219724
- [Derived] Shahidi N, Vosko S, Gupta S, van Hattem WA, Sidhu M, Tate DJ, Williams SJ, Lee EYT, Burgess N, Bourke MJ. Previously Attempted Large Nonpedunculated Colorectal Polyps Are Effectively Managed by Endoscopic Mucosal Resection. Am J Gastroenterol. 2021 May 1;116(5):958-966. doi: 10.14309/ajg.0000000000001096. PMID 33625125
- [Derived] Tate DJ, Sidhu M, Bar-Yishay I, Desomer L, Brown G, Hourigan LF, Lee EYT, Moss A, Raftopoulos S, Singh R, Williams SJ, Zanati S, Burgess N, Bourke MJ. Impact of en bloc resection on long-term outcomes after endoscopic mucosal resection: a matched cohort study. Gastrointest Endosc. 2020 May;91(5):1155-1163.e1. doi: 10.1016/j.gie.2019.12.025. Epub 2019 Dec 28. PMID 31887274
- [Derived] Tate DJ, Desomer L, Hourigan LF, Moss A, Singh R, Bourke MJ. Two-stage endoscopic mucosal resection is a safe and effective salvage therapy after a failed single-session approach. Endoscopy. 2017 Sep;49(9):888-898. doi: 10.1055/s-0043-110671. Epub 2017 May 31. PMID 28564715
- [Derived] Tate DJ, Desomer L, Klein A, Brown G, Hourigan LF, Lee EY, Moss A, Ormonde D, Raftopoulos S, Singh R, Williams SJ, Zanati S, Byth K, Bourke MJ. Adenoma recurrence after piecemeal colonic EMR is predictable: the Sydney EMR recurrence tool. Gastrointest Endosc. 2017 Mar;85(3):647-656.e6. doi: 10.1016/j.gie.2016.11.027. Epub 2016 Nov 28. PMID 27908600
- [Derived] Burgess NG, Bassan MS, McLeod D, Williams SJ, Byth K, Bourke MJ. Deep mural injury and perforation after colonic endoscopic mucosal resection: a new classification and analysis of risk factors. Gut. 2017 Oct;66(10):1779-1789. doi: 10.1136/gutjnl-2015-309848. Epub 2016 Jul 27. PMID 27464708
- [Derived] Bahin FF, Rasouli KN, Williams SJ, Lee EY, Bourke MJ. Prophylactic clipping for the prevention of bleeding following wide-field endoscopic mucosal resection of laterally spreading colorectal lesions: an economic modeling study. Endoscopy. 2016 Aug;48(8):754-61. doi: 10.1055/s-0042-105558. Epub 2016 Apr 25. PMID 27110693
- [Derived] Tutticci N, Klein A, Sonson R, Bourke MJ. Endoscopic resection of subtotal or completely circumferential laterally spreading colonic adenomas: technique, caveats, and outcomes. Endoscopy. 2016 May;48(5):465-71. doi: 10.1055/s-0042-101854. Epub 2016 Mar 23. PMID 27009082
- [Derived] Pellise M, Burgess NG, Tutticci N, Hourigan LF, Zanati SA, Brown GJ, Singh R, Williams SJ, Raftopoulos SC, Ormonde D, Moss A, Byth K, P'Ng H, Mahajan H, McLeod D, Bourke MJ. Endoscopic mucosal resection for large serrated lesions in comparison with adenomas: a prospective multicentre study of 2000 lesions. Gut. 2017 Apr;66(4):644-653. doi: 10.1136/gutjnl-2015-310249. Epub 2016 Jan 19. PMID 26786685
- [Derived] Pellise M, Desomer L, Burgess NG, Williams SJ, Sonson R, McLeod D, Bourke MJ. The influence of clips on scars after EMR: clip artifact. Gastrointest Endosc. 2016 Mar;83(3):608-16. doi: 10.1016/j.gie.2015.08.071. Epub 2015 Sep 10. PMID 26364966
- [Derived] Jayanna M, Burgess NG, Singh R, Hourigan LF, Brown GJ, Zanati SA, Moss A, Lim J, Sonson R, Williams SJ, Bourke MJ. Cost Analysis of Endoscopic Mucosal Resection vs Surgery for Large Laterally Spreading Colorectal Lesions. Clin Gastroenterol Hepatol. 2016 Feb;14(2):271-8.e1-2. doi: 10.1016/j.cgh.2015.08.037. Epub 2015 Sep 11. PMID 26364679
- [Derived] Nanda KS, Tutticci N, Burgess NG, Sonson R, Williams SJ, Bourke MJ. Endoscopic mucosal resection of laterally spreading lesions involving the ileocecal valve: technique, risk factors for failure, and outcomes. Endoscopy. 2015 Aug;47(8):710-8. doi: 10.1055/s-0034-1391732. Epub 2015 Mar 12. PMID 25763831
- [Derived] Burgess NG, Pellise M, Nanda KS, Hourigan LF, Zanati SA, Brown GJ, Singh R, Williams SJ, Raftopoulos SC, Ormonde D, Moss A, Byth K, P'Ng H, McLeod D, Bourke MJ. Clinical and endoscopic predictors of cytological dysplasia or cancer in a prospective multicentre study of large sessile serrated adenomas/polyps. Gut. 2016 Mar;65(3):437-46. doi: 10.1136/gutjnl-2014-308603. Epub 2015 Mar 2. PMID 25731869
- [Derived] Moss A, Williams SJ, Hourigan LF, Brown G, Tam W, Singh R, Zanati S, Burgess NG, Sonson R, Byth K, Bourke MJ. Long-term adenoma recurrence following wide-field endoscopic mucosal resection (WF-EMR) for advanced colonic mucosal neoplasia is infrequent: results and risk factors in 1000 cases from the Australian Colonic EMR (ACE) study. Gut. 2015 Jan;64(1):57-65. doi: 10.1136/gutjnl-2013-305516. Epub 2014 Jul 1. PMID 24986245